CLINICAL TRIAL: NCT02475148
Title: A Randomized, Placebo-controlled, Double-blind, Single Ascending Dose Study to Investigate Safety and Tolerability, Pharmacokinetics, Pharmacodynamics and Food Effect of JNJ-54175446 in Healthy Subjects
Brief Title: A Study to Investigate Safety and Tolerability, Pharmacokinetics, Pharmacodynamics and Food Effect of JNJ-54175446 in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen-Cilag International NV (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR107482; 2015-000942-53 (EudraCT Number); 54175446EDI1001 (Other: Janssen-Cilag International NV)
Record Dates: First submitted 2015-06-16; First posted 2015-06-18 (Estimated); Last update posted 2025-02-03 (Actual); Status verified 2025-01

CONDITIONS: Healthy
Keywords: JNJ-54175446; Healthy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (8):
- Part 1: Cohort 1 (Experimental): Participants will receive either JNJ-54175446 0.5 milligram (mg) or placebo on Day 1.
  Interventions: Drug: JNJ 54175446; Drug: Placebo
- Part 1: Cohort 2 (Experimental): Participants will receive either JNJ-54175446 2.5 mg or placebo on Day 1.
  Interventions: Drug: JNJ 54175446; Drug: Placebo
- Part 1: Cohort 3 (Experimental): Participants will receive either JNJ-54175446 10 mg or placebo on Day 1.
  Interventions: Drug: JNJ 54175446; Drug: Placebo
- Part 1: Cohort 4 (Experimental): Participants will receive either JNJ-54175446 30 mg or placebo on Day 1.
  Interventions: Drug: JNJ 54175446; Drug: Placebo
- Part 1: Cohort 5 (Experimental): Participants will receive either JNJ-54175446 100 mg or placebo on Day 1.
  Interventions: Drug: JNJ 54175446; Drug: Placebo
- Part 1: Cohort 6 (Experimental): Participants will receive either JNJ-54175446 200 mg or placebo on Day 1.
  Interventions: Drug: JNJ 54175446; Drug: Placebo
- Part 2: Cohort 7 (Experimental): Participants will receive JNJ-54175446 on Day 1. The dose of JNJ-54175446 will be determined in part 1 as suitable dose.
  Interventions: Drug: JNJ 54175446
- Part 3: Cohort 8 (Experimental): Participants will receive JNJ-54175446 on Day 1 along with high fat/high calorie breakfast. The dose of JNJ-54175446 will be determined in part 1 as suitable dose.
  Interventions: Drug: JNJ 54175446; Drug: Placebo; Other: High fat/high Calorie Breakfast

INTERVENTIONS:
Drug: JNJ 54175446
Drug: Placebo
  Arms: Part 1: Cohort 1; Part 1: Cohort 2; Part 1: Cohort 3; Part 1: Cohort 4; Part 1: Cohort 5; Part 1: Cohort 6; Part 3: Cohort 8
Other: High fat/high Calorie Breakfast
  Arms: Part 3: Cohort 8

SUMMARY:
The purpose of this study is to investigate the safety and tolerability of JNJ-54175446 versus placebo after single oral dose administration (ascending dose levels), to determine the maximal tolerated dose (MTD) or the safety and tolerability at exposures resulting in full target engagement for at least 24 hours in all participants (whichever comes first), to characterize the pharmacokinetics of JNJ-54175446 in plasma, cerebrospinal fluid (CSF) and urine and to investigate the effect of food (high fat/high calorie) on the pharmacokinetics of JNJ 54175446 after single oral dose administration.

DETAILED DESCRIPTION:
This is a double-blind, placebo-controlled, randomized, single ascending dose study in healthy participants for JNJ-54175446. The study will consist of 3 phases: a screening phase (between 21 and 2 days prior to dose administration), a double-blind treatment phase (8 days; Part 1 and Part 3) or an open-label treatment phase (8 days; Part 2), and a follow-up examination (within 14 to 21 days after dose administration). The maximal study duration for a participant will not exceed 6 weeks. In each cohort of Part 1 (6 cohorts) and Part 3 (1 cohort), participants will be randomly assigned to receive JNJ-54175446 or matching placebo and in cohort of part 2, all participants will be assigned to JNJ-54175446 treatment. In part 1, primarily maximum tolerated dose (MTD) will be assessed, along with safety and tolerability of JNJ-54175446. In part 2, pharmacokinetics (PK) of JNJ-54175446 in cerebrospinal fluid (CSF) will be assessed. In part 3, the effect of food on the plasma PK of JNJ-54175446 in young healthy male participants will be assessed. Safety will be monitored throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have a body mass index (BMI) between 18 and 32 kg/m^2, inclusive (BMI = weight/height^2)
* Participants must be healthy on the basis of clinical laboratory tests performed at screening. If the results of the serum chemistry panel[excluding liver function tests], hematology, or urinalysis are outside the normal reference ranges, the participant may be included only if the investigator judges the abnormalities to be not clinically significant. This determination must be recorded in the subject's source documents and initialed by the investigator
* A man who is sexually active with a woman of childbearing potential and has not had a vasectomy must agree to use a barrier method of birth control e.g., either condom with spermicidal foam/gel/film/cream/suppository or partner with occlusive cap (diaphragm or cervical/vault caps) with spermicidal foam/gel/film/cream/suppository, and all men must also not donate sperm during the study and for 3 months after receiving the last dose of study drug. In addition, their female partner should also use an appropriate method of birth control for at least the same duration

For Part 1 and 3:

- Healthy male participants between 18 and 54 years of age, inclusive

For Part 2:

* Healthy male or female participants between 55 and 75 years of age, inclusive
* Participant must be healthy on the basis of both physical and neurological examination performed at screening and at admission to the clinical unit
* Women must not be of childbearing potential (i.e., must be postmenopausal with amenorrhea for at least 12 months); permanently sterilized (e.g., tubal occlusion, hysterectomy, bilateral salpingectomy); or otherwise be incapable of pregnancy

Exclusion Criteria:

* Participant has a history of or current liver or renal insufficiency; significant cardiac, vascular, pulmonary, gastrointestinal, endocrine, neurologic, hematologic (including coagulation disorders), rheumatologic, psychiatric, or metabolic disturbances, any inflammatory illness or any other illness that the Investigator considers should exclude the participant
* Participant has any liver function test (including alanine aminotransferase [ALT], aspartate aminotransferase [AST], gamma-glutamyltransferase [gamma-GT], alkaline phosphatase [ALP] and bilirubin) at screening exceeding the upper limit of normal
* Participant has a history of hepatitis B surface antigen (HBsAg) or hepatitis C antibody (anti-HCV) positive, or other clinically active liver disease, or tests positive for HBsAg or anti-HCV at Screening
* Participant has a history of human immunodeficiency virus (HIV) antibody positive, or tests positive for HIV at Screening
* Participant has a Prothrombin time [PT] >14 seconds and/or an activated partial thromboplastin time [aPTT] >35 seconds

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2015-06; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Adverse Events | Baseline up to 14 or 21 days after study drug administration
  An adverse event is any untoward medical event that occurs in a participant administered an investigational product, and it does not necessarily indicate only events with clear causal relationship with the relevant investigational product.
Maximum Tolerated Dose of JNJ-54175446 in Part 1 | Baseline up to 24 Hours after study drug administration
Maximum Observed Plasma and Cerebrospinal Fluid (CSF) Concentration (Cmax) | Pre-dose; 0.5, 1, 1.5, 2, 3, 4, 6, 9, 12, 18, 24, 36, 48, 72, 96, 120, 144 hours after study drug administration
  The Cmax is the maximum observed concentration.
Last Quantifiable Plasma and Cerebrospinal Fluid (CSF) Concentration (Clast) | Pre-dose; 0.5, 1, 1.5, 2, 3, 4, 6, 9, 12, 18, 24, 36, 48, 72, 96, 120, 144 hours after study drug administration
Time to Reach Maximum Observed Plasma and Cerebrospinal Fluid Concentration (Tmax) | Pre-dose; 0.5, 1, 1.5, 2, 3, 4, 6, 9, 12, 18, 24, 36, 48, 72, 96, 120, 144 hours after study drug administration
Time to Last Quantifiable Plasma and Cerebrospinal Fluid Concentration (Tlast) | Pre-dose; 0.5, 1, 1.5, 2, 3, 4, 6, 9, 12, 18, 24, 36, 48, 72, 96, 120, 144 hours after study drug administration
Area Under Curve From Time of Administration up to the Last Time Point with a Measurable Plasma and Cerebrospinal Fluid Concentration (AUClast) | Pre-dose; 0.5, 1, 1.5, 2, 3, 4, 6, 9, 12, 18, 24, 36, 48, 72, 96, 120, 144 hours after study drug administration
Area Under the Plasma and Cerebrospinal Fluid Concentration-Time Curve From Time Zero to Infinite Time (AUC[0-infinity]) | Pre-dose; 0.5, 1, 1.5, 2, 3, 4, 6, 9, 12, 18, 24, 36, 48, 72, 96, 120, 144 hours after study drug administration
First-order Rate Constant (Lambda[z]) | Pre-dose; 0.5, 1, 1.5, 2, 3, 4, 6, 9, 12, 18, 24, 36, 48, 72, 96, 120, 144 hours after study drug administration
Elimination Half-Life (t1/2) | Pre-dose; 0.5, 1, 1.5, 2, 3, 4, 6, 9, 12, 18, 24, 36, 48, 72, 96, 120, 144 hours after study drug administration
  The elimination half-life (t1/2) is the time measured for the plasma/CSF concentration to decrease by 1 half to its original concentration. It is associated with the terminal slope of the semi logarithmic drug concentration-time curve, and is calculated as 0.693/lambda(z).
Total Clearance (CL/F) | Pre-dose; 0.5, 1, 1.5, 2, 3, 4, 6, 9, 12, 18, 24, 36, 48, 72, 96, 120, 144 hours after study drug administration
  Total clearance of drug after extravascular administration, uncorrected for absolute bioavailability
Creatinine Clearance | Pre-dose; 0.5, 1, 1.5, 2, 3, 4, 6, 9, 12, 18, 24, 36, 48, 72, 96, 120, 144 hours after study drug administration
  Creatinine clearance was calculated by Cockroft-Gault formula. Creatinine clearance is equal to 140 minus age multiplied by weight and constant (1 for men and 0.85 for women) divided by creatinine in (micro mole per liter).

CONTACTS AND LOCATIONS:
Overall Officials: Janssen-Cilag International NV Clinical Trial, Study Director — Janssen-Cilag International NV
Locations (1):
- Merksem, Belgium

REFERENCES:
- [Derived] Triana-Baltzer G, Timmers M, De Boer P, Schoene M, Furey M, Bleys C, Vrancken I, Slemmon R, Ceusters M, van Nueten L, Kolb H. Profiling classical neuropsychiatric biomarkers across biological fluids and following continuous lumbar puncture: A guide to sample type and time. Compr Psychoneuroendocrinol. 2022 Jan 15;10:100116. doi: 10.1016/j.cpnec.2022.100116. eCollection 2022 May. PMID 35774109